CLINICAL TRIAL: NCT04917679
Title: Eltrombopag Plus Diacerein vs Eltrombopag in Adult Primary Immune Thrombocytopenia: a Multicenter Randomized Controlled Trial
Brief Title: Eltrombopag Plus Diacerein vs Eltrombopag in Adult ITP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eltrombopag-Diacerein ITP
Record Dates: First submitted 2020-12-01; First posted 2021-06-08 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-06

CONDITIONS: Thrombocytopenia
Keywords: ITP; Eltrombopag; Diacerein
MeSH Terms: conditions — Thrombocytopenia | interventions — eltrombopag; diacerein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination group (Experimental): Eltrombopag plus diacerein
  Interventions: Drug: Eltrombopag plus diacerein
- Monotherapy group (Placebo Comparator): Eltrombopag monotherapy
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag plus diacerein — In the combination group, eltrombopag will be administered orally at an initial dose of 75mg daily for 14 days, and diacerein will be given orally at an initial dose of 50mg bid concomitantly for 14 days (D1-D14). During treatment period, treating physicians will modify the dosage of trial treatment to maintain participants' platelet count at the range of 50 - 150 × 10^9/L as follows: (1) if platelet count is less than 150 × 10^9/L, continue the original treatment (eltrombopag 75mg daily plus diacerein 50mg bid); (2) if platelet count is between 150 × 10^9/L to 250 × 10^9/L, the treatment will be modified to eltrombopag 50mg daily plus diacerein 50mg bid; (3) if platelet count is over 250 × 10^9/L, original treatment (both eltrombopag and diacerein) need to be stopped, and platelet count should be reexamined every other day, and the treatment (eltrombopag 50mg daily plus diacerein 50mg bid ) will be restarted until platelet count is below 100 × 10^9/L.
  Arms: Combination group
Drug: Eltrombopag — In the monotherapy group, eltrombopag also will be administered orally at an initial dose of 75mg daily for 14 days (D1-D14), and the individualized dosage could be modified by treating physicians to maintain participants' platelet count between 50 × 10^9/L to 150 × 10^9/L.
  Arms: Monotherapy group

SUMMARY:
Primary immune thrombocytopenia (ITP) is an autoimmune bleeding disorder with low platelet count. As the first choice of the second-line treatment of ITP, thrombopoietin receptor agonist (TPO-RA) enable long-term remission in 50% to 60% of cases. However, about half of patients have no response or loss of response to eltrombopag due to unknown reasons, which can't be effectively improved by increasing the drug dose. Diacerein is an anthraquinone derivative used to treat joint diseases such as osteoarthritis. We speculate that the addition of diacerein to eltrombopag may offer sensitizer effect and maximize efficacy, which warrants further prospective studies to evaluate the efficacy and safety of the combination therapy as salvage strategy in ameliorating immune thrombocytopenia.

DETAILED DESCRIPTION:
In this multicentre, open-label, randomized controlled trial, 98 eltrombopag-inefficient or relapsed ITP patients will be enrolled from five tertiary medical centres in China. Participants will be randomly assigned into the combination group (eltrombopag orally at initial dose of 75 mg daily for 14 days, plus diacerein orally at initial dose of 50 mg bid for 14 days) or the monotherapy group (eltrombopag orally at initial dose of 75 mg daily for 14 days) by masked statisticians in a 1:1 ratio. The primary endpoints are initial response at D15 without any additional ITP-specific intervention. The secondary outcomes include response at D28, time to response, duration of response, bleeding score, health-related quality of life assessment, and safety issue. This study will compare the efficacy and safety of eltrombopag-diacerein with eltrombopag monotherapy in adults with primary immune thrombocytopenia. We hypothesized that the novel combination of eltrombopag and diacerein might extend eltrombopag efficacy and avoid rapid alteration to less-preferable therapies, especially in the management of the patient refractory to eltrombopag.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age at the time of the screening.
* Participant may be male or female.
* Participant has a confirmed diagnosis of ITP according to the 2019 International Working Group assessment at screening.
* Participant who didn't respond to eltrombopag retreatment (75mg by mouth once a day for 14 days) after eltrombopag previous treatment inefficient or relapsed (platelet count below 30 × 10^9/L or below 2-fold increase from baseline platelet count, or bleeding).
* Bone marrow biopsy is performed in participants over 60 years to exclude hematological malignancies.

Exclusion Criteria:

* Participant has evidence of a secondary cause of immune thrombocytopenia (e.g. leukemia, lymphoma, common variable immune-deficiency, systemic lupus erythematosus, autoimmune thyroid disease, past medical history of untreated H. pylori infection) or to drug treatments (e.g. heparin, quinine, antimicrobials, anticonvulsants) or participant has a multiple immune cytopenia, e.g. Evan's syndrome.
* Participant has clinically life-threatening bleeding (e.g. central nervous system bleeding, menorrhagia with significant drop in hemoglobin). Participant has a history of coagulopathy disorders other than ITP.
* Participant has a history of arterial or venous thromboembolism (e.g. stroke, transient ischemic attach, myocardial infarction, deep vein thrombosis or pulmonary embolism) within the 6 months prior to randomization or requires anticoagulant treatment.
* Participant has 12-lead ECG with changes considered to be clinically significant upon medical review at baseline.
* Participant has severe renal impairment (glomerular filtration rate less than 45ml/min/1.73 m2).
* Participant has 3 × upper limit of normal of any of the following: alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase.
* Participant has received corticosteroids, rh-TPO, romiplostim, or immunosuppression within 4 weeks before screening.
* Participant with any of the following conditions: severe immunodeficiency, active or previous malignancy, human immunodeficiency virus (HIV), hepatitis B or C virus infection, pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Initial response at Day 15 | Day 15
  The primary outcomes of this trial are initial responses at Day 15 without any additional ITP-specific intervention. Complete response was defined as a platelet count at or above 100 × 10⁹ cells per L and an absence of bleeding. Partial response was defined as a platelet count at or above 30 × 10⁹ cells per L but less than 100 × 10⁹ cells per L and at least a doubling of the baseline platelet count and an absence of bleeding. No response was defined as a platelet count of less than 30 × 10⁹ cells per L, or less than two-times increase from baseline platelet count, or bleeding.

SECONDARY OUTCOMES:
Response at Day 28 | Day 28
  Responses were assessed at day 28. Complete response was defined as a platelet count at or above 100 × 10⁹ cells per L and an absence of bleeding. Partial response was defined as a platelet count at or above 30 × 10⁹ cells per L but less than 100 × 10⁹ cells per L and at least a doubling of the baseline platelet count and an absence of bleeding. No response was defined as a platelet count of less than 30 × 10⁹ cells per L, or less than two-times increase from baseline platelet count, or bleeding.
Time to response | 28 days
  Time to response was defined as the time from treatment initiation to achieve a complete response or a partial response, whichever came first, assessed up to day 28.
Duration of response | 12 months
  Duration of response was defined as the time from achievement of a complete response or a partial response to the loss of response (platelet count <30 × 10⁹ cells per L; measured on two occasions more than 1 day apart or the presence of bleeding).
Bleeding scores | 12 months
  Bleeding symptoms were graded according a standardized bleeding scale specific to primary immune thrombocytopenia on the basis of site and severity of bleeding by Khellaf et al (PMID: 15951296). A modification was made to exclude age from the original scale so that only bleeding symptoms were described. At each visit, we recorded bleeding scores. Routine visits were scheduled once a week for the first 4 weeks and once a month thereafter. Scores ranged from 0 to 59, with higher values indicating higher bleeding risk.
Health-related quality of life assessment | 12 weeks
  Health-related quality of life was assessed using a self-administered immune thrombocytopenia Patient Assessment Questionnaire (ITP-PAQ) at baseline and at week 12. Scores ranged from 0 to 100, with higher values indicating better quality of life.
The number of participants with Adverse events | 12 months
  Adverse events were graded according to the Common Terminology Criteria for Adverse Events (version 4.0). At each visit, we recorded adverse events. Routine visits were scheduled once a week for the first 4 weeks and once a month thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hou, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Derived] Sun L, Huang X, Wang J, Yuan C, Zhao H, Li D, Xu R, Wang Y, Qin P, Shi Y, Peng J, Hou M, Hou Y. Eltrombopag plus diacerein vs eltrombopag in patients with ITP: a multicenter, randomized, open-label phase 2 trial. Blood. 2024 Oct 24;144(17):1791-1799. doi: 10.1182/blood.2024025067. PMID 38958479